CLINICAL TRIAL: NCT04028063
Title: An Open-Label, Phase II Efficacy Trial of Doxorubicin in Combination With Dual Checkpoint Blockade Using Zalifrelimab (AGEN1884) or Botensilimab (AGEN1181) With Balstilimab (AGEN2034) for Advanced or Metastatic Soft Tissue Sarcomas
Brief Title: Doxorubicin Plus Dual Checkpoint Blockade for Soft Tissue Sarcomas
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Agenus Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 19-0554.cc; NCI-2020-00728 (Other: CTRP)
Record Dates: First submitted 2019-07-17; First posted 2019-07-22 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Soft Tissue Sarcoma; Advanced Soft Tissue Sarcoma
MeSH Terms: conditions — Sarcoma | interventions — balstilimab; Doxorubicin; liposomal doxorubicin

STUDY DESIGN:
Intervention Model Description: This is an open-label, non-randomized, single-institution, single arm Phase II study conducted using a Simon two-stage design with an additional safety lead-in.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Part 1: Stage 1, Safety Lead-In (Experimental): The safety lead-in will enroll 6 participants. Balstilimab 300mg flat q3 weeks up to 2 years; Zalifrelimab 1mg/kg q6 weeks x 4; Doxorubicin 75mg/m2 q3 weeks x 2, starts at C2 The participants will complete a dose-limiting toxiciy (DLT) observation period of 9 weeks.
  Interventions: Drug: Balstilimab; Drug: Zalifrelimab; Drug: Doxorubicin
- Part 1: Stage 2, Expansion (Experimental): Balstilimab 300mg flat q3 weeks up to 2 years; Zalifrelimab 1mg/kg q6 weeks up to 2 years; Doxorubicin 75mg/m2 q3 weeks x 6
  Interventions: Drug: Balstilimab; Drug: Zalifrelimab; Drug: Doxorubicin
- Part 2: Stage 2, Dose 1 (Experimental): Doxorubicin 60mg/m2 q3 weeks x 6 doses Botensilimab 75mg q6 weeks up to two years
  Interventions: Drug: Doxorubicin; Drug: Botensilimab
- Stage 2, Dose 2 (Experimental): Doxorubicin 75mg/m2 q3 weeks x 6 doses Botensilimab 75mg q6 weeks up to two years
  Interventions: Drug: Doxorubicin; Drug: Botensilimab
- Stage 2, Dose 3 Combination of Doxorubicin with Botensilimab and Balstilimab (Experimental): Doxorubicin 75mg/m2 q3 weeks x 6 doses Botensilimab 75mg flat q6 weeks up to 2 years Balstilimab 450mg q3 weeks up to 2 years
  Interventions: Drug: Balstilimab; Drug: Doxorubicin; Drug: Botensilimab

INTERVENTIONS:
Drug: Balstilimab — Balstilimab (AGEN2034) is a human monoclonal antibody that targets programmed cell death 1 (PD-1). Engagement of PD-1 by its ligands, programmed death ligand (PD-L1) and PD-L2, leads to signal transduction that inhibits important aspects of T cell function including proliferation, cytokine production and cytolytic activity. Balstilimab (AGEN2034) potently inhibits PD-1 binding to PD- L1 and PD- L2 and is intended to reverse the immunosuppressive effects of this signaling pathway in the context of tumor immuno-surveillance by T cells. Balstilimab (AGEN2034) is intended for development as a treatment for advanced malignancies as a single agent or in combinations.
  Other Names: AGEN2034
  Arms: Part 1: Stage 1, Safety Lead-In; Part 1: Stage 2, Expansion; Stage 2, Dose 3 Combination of Doxorubicin with Botensilimab and Balstilimab
Drug: Zalifrelimab — Zalifrelimab (AGEN1884) is a fully human monoclonal immunoglobulin G1 κ subclass (IgG1κ) antibody that specifically recognizes cytotoxic T lymphocyte-associated protein 4 (CTLA-4, also known as CD152). Zalifrelimab (AGEN1884) is being developed as a monotherapy for cancer indications with potential for future development in combination with other immunotherapies.
  Other Names: AGEN1884
  Arms: Part 1: Stage 1, Safety Lead-In; Part 1: Stage 2, Expansion
Drug: Doxorubicin — Doxorubicin is the standard of care first-line therapy for most subtypes of metastatic soft tissue sarcomas. Doxorubicin monotherapy administered at 75 mg/m2 has resulted in objective response rate of 14%, and median progression-free survival of 4.6 months, and another study reported progression-free survival at 6 months of 46.3%, with a median PFS of 5.8 months, and best objective response rate of 19%.
  Other Names: Lipodox, Doxil
Drug: Botensilimab — Botensilimab (AGEN1181) is a novel, human, fragment-crystallizable (Fc)-engineered immunoglobulin G1 (IgG1) anti-CTLA-4 antibody designed to exploit a novel mechanism by which increased Fc engagement enhances antigen-specific effector T cell responses.
  Other Names: AGEN1181
  Arms: Part 2: Stage 2, Dose 1; Stage 2, Dose 2; Stage 2, Dose 3 Combination of Doxorubicin with Botensilimab and Balstilimab

SUMMARY:
This is an open-label, non-randomized, single-institution, single arm Phase II study conducted using a Simon two-stage design with an additional safety lead-in. The overall objective is to determine the efficacy of combination doxorubicin with dual checkpoint blockade with anti-CTLA-4 antibody AGEN1884 and anti-PD-1 antibody AGEN2034. The investigators will estimate the progression-free survival rate at 6 months (PFS6mo) of doxorubicin plus AGEN1884/AGEN2034 in comparison to historical PFS6mo with doxorubicin monotherapy, calculated as the mean from two large randomized Phase 3 clinical trials.

DETAILED DESCRIPTION:
The primary endpoint for the study is PFS6mo by RECIST 1.1. The sample size calculation is based on a Simon Two-Stage design with incorporation of early stopping rules for safety and futility (See section 9 for statistical considerations). The Investigators will enroll up to 35 patients on the study to obtain 28 evaluable patients for the primary endpoint. Safety of the combination will be evaluated after the first six patients complete the DLT observation period of 9 weeks. This lengthy DLT period is designed to capture safety and toxicity profile, understanding that immune-related toxicities from checkpoint inhibitors may not emerge immediately. This will also ensure adequate evaluation of potential cardiac and hepatic toxicity from combination doxorubicin and checkpoint inhibitor therapy. If two or more patients experience DLT in the initial safety lead-in cohort, the regimen will be declared intolerable. Any patients who do not complete study therapy through the 9-week DLT observation period for any reasons other than toxicity will be replaced for safety lead-in assessment. If fewer than two patients experience DLT, the investigators will proceed to expansion to complete enrollment of 15 patients in Stage 1. Following enrollment of stage one, accrual will pause for analysis of efficacy. If 6 or fewer of the 15 patients are progression-free at 6 months, the investigators will halt the study for futility. If 7 or more patients are free from progression, then the investigators will proceed with enrollment of 13 additional patients to complete stage 2. the investigators are powered to detect improvement in 6-month PFS rate to 63.4% with the combination over the 43.4% historical PFS6mo.

ELIGIBILITY:
Inclusion Criteria:

Part One:

1. Provision to sign and date the consent form.
2. Stated willingness to comply with all study procedures and be available for the duration of the study.
3. Be male or female aged 18-100 years at the time of signing informed consent.
4. Have a histological diagnosis of advanced or metastatic soft tissue sarcoma (STS) (by local pathology review), not curable by surgery, for which treatment with doxorubicin is deemed appropriate by the investigator.
5. Has one of the following histologies:

   * synovial sarcoma,
   * malignant peripheral nerve sheath tumors,
   * dedifferentiated, pleomorphic or myxoid/round cell liposarcoma,
   * uterine or soft tissue leiomyosarcoma,
   * malignant phylloides tumor,
   * high grade undifferentiated pleomorphic sarcomas (HGUPS/MFH),
   * myxofibrosarcoma,
   * fibrosarcoma,
   * angiosarcoma,
   * spindle cell or undifferentiated sarcoma NOS,
   * malignant myoepithelioma,
   * malignant solitary fibrous tumor/hemangiopericytoma,
   * epithelioid hemangioendothelioma,
   * Any other histology or standard of care treatment not specifically addressed will be reviewed by the principal investigator and pathologist for final determination of eligibility.
6. Have measurable or nonmeasurable but evaluable disease as defined by the Response Evaluation Criteria in Solid Tumors (RECIST 1.1). Tumors within a previously irradiated field will be designated as "nontarget" lesions unless progression is documented or a biopsy is obtained to confirm persistence at least 90 days following completion of radiotherapy.
7. Have received 0 or 1 prior systemic therapies for metastatic sarcoma and NO prior anthracyclines or checkpoint inhibitors.
8. Adequate organ function as defined in protocol.

   Absolute neutrophil count (ANC) ≥1,000 /mcL Platelets ≥100,000 / mcL Hemoglobin ≥8 g/dL without EPO dependency

   Serum creatinine OR Measured or calculated creatiniecclearance

   ≤1.5 X upper limit of normal (ULN) OR ≥60 mL/min for subject with creatinine levels > 1.5 X institutional ULN

   Serum total bilirubin ≤ 1.5 X ULN OR Direct bilirubin ≤ ULN for subjects with total bilirubin levels > 1.5 ULN Exception: Subjects with known history of Gilbert's disease should be ≤ 1.5 X of the patient's prior baseline AST (SGOT) and ALT (SGPT) ≤2.5 X ULN OR ≤ 5 X ULN for subjects with liver metastases Albumin >2.5 mg/dL

   International Normalized Ratio (INR) or Prothrombin Time (PT)

   ≤1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants

   Activated Partial Thromboplastin Time (aPTT) ≤1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants

   Creatinine clearance should be calculated per institutional standard.
9. ECOG performance status of 0 or 1.
10. Patients must consent and be willing to undergo tumor core needle biopsies at two timepoints: 1. Baseline, 2. Cycle 2 Day 5; a third biopsy for off-study/progression is optional but advised. At least one tumor site must be amenable to biopsy in the judgment of the interventional radiologist.
11. Female subjects of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
12. Females of child bearing potential that are sexually active must agree to either practice 2 medically accepted highly effective methods of contraception at the same time or abstain from heterosexual intercourse from the time of signing the informed consent through 120 days after the last dose of study drug. See Appendix B for protocol-approved highly effective methods of contraceptive combinations. Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.

    * Negative test for pregnancy is required of females of child-bearing potential. A female of child-bearing potential is any woman, regardless of sexual orientation or whether they have undergone tubal ligation, who meets the following criteria: 1. Has not undergone a hysterectomy or bilateral oophorectomy; or 2. Has not been naturally postmenopausal for at least 24 consecutive months (ie, has had menses at any time in the preceding 24 consecutive months or 730 days.)
    * Conception while on treatment must be avoided.
13. Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy. Prior history of vasectomy does NOT replace requirement for contraceptive use.
14. Subjects must either possess or undergo placement of central venous catheter, including pheresis or trifusion catheter, PICC line, or port.

Part Two: In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. Provision to sign and date the consent form.
2. Stated willingness to comply with all study procedures and be available for the duration of the study.
3. Be male or female aged 18-100 years at the time of signing informed consent.
4. Have a histological diagnosis of advanced or metastatic soft tissue sarcoma (STS) (by local pathology review), not curable by surgery, for which treatment with doxorubicin is deemed appropriate by the investigator.
5. Has one of the following histologies:

   * synovial sarcoma,
   * malignant peripheral nerve sheath tumors,
   * dedifferentiated, pleomorphic or myxoid/round cell liposarcoma,
   * uterine or soft tissue leiomyosarcoma,
   * malignant phylloides tumor,
   * high grade undifferentiated pleomorphic sarcomas (HGUPS/MFH),
   * myxofibrosarcoma,
   * fibrosarcoma,
   * angiosarcoma,
   * spindle cell or undifferentiated sarcoma NOS,
   * malignant myoepithelioma,
   * malignant solitary fibrous tumor/hemangiopericytoma,
   * epithelioid hemangioendothelioma,
   * Any other histology or standard of care treatment not specifically addressed will be reviewed by the principal investigator in consultation with pathology as needed for final determination of eligibility.
6. Have measurable or nonmeasurable but evaluable disease as defined by the Response Evaluation Criteria in Solid Tumors (modified RECIST 1.1). Tumors within a previously irradiated field will be designated as "nontarget" lesions unless progression is documented or a biopsy is obtained to confirm persistence at least 90 days following completion of radiotherapy.
7. Have received any number of prior systemic therapies for metastatic sarcoma but NO prior anthracyclines or checkpoint inhibitors. Re-treatment with the same drug or regimen after interruption (i.e. chemotherapy holiday) is not considered a new line of treatment, and those patients are eligible.
8. Adequate organ function as defined in protocol.

   Absolute neutrophil count (ANC) ≥1,000 /mcL Platelets ≥100,000 / mcL Hemoglobin ≥8 g/dL without EPO dependency

   Serum creatinine OR Measured or calculated creatinine clearance (GFR can also be used in place of creatinine or CrCl)

   ≤1.5 X upper limit of normal (ULN) OR ≥60 mL/min for subject with creatinine levels > 1.5 X institutional ULN

   Serum total bilirubin ≤ 1.5 X ULN OR Direct bilirubin ≤ ULN for subjects with total bilirubin levels > 1.5 ULN. Exception: Subjects with known history of Gilbert's disease should be ≤ 1.5 X of the patient's prior baseline

   AST (SGOT) and ALT (SGPT) ≤ 2.5 X ULN OR ≤ 5 X ULN for subjects with liver metastases Albumin >2.5 mg/dL

   International Normalized Ratio (INR) or Prothrombin Time (PT) ≤1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants

   Activated Partial Thromboplastin Time (aPTT) ≤1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants Creatinine clearance should be calculated per institutional standard.
9. ECOG performance status of 0 or 1.
10. Patients must consent and be willing to undergo tumor core needle biopsies at two timepoints: 1. Baseline, 2. Cycle 2 Day 5; a third biopsy for off-study/progression is optional but advised. At least one tumor site must be amenable to biopsy in the judgment of the investigator, with consultation with the interventional radiologist as needed.
11. Female subjects of childbearing potential must have a negative urine or serum pregnancy test at screening. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required. In the rare case where the sarcoma is thought to be producing beta HCG, patients with a positive serum HCG test must have a uterine ultrasound for confirmation of negative pregnancy status.
12. Females of child bearing potential that are sexually active must agree to either practice 2 medically accepted highly effective methods of contraception at the same time or abstain from heterosexual intercourse from the time of signing the informed consent through 120 days after the last dose of study drug. See Appendix B for protocol-approved highly effective methods of contraceptive combinations. Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.

    * Negative test for pregnancy is required of females of child-bearing potential. A female of child-bearing potential is any woman, regardless of sexual orientation or whether they have undergone tubal ligation, who meets the following criteria: 1. Has not undergone a hysterectomy or bilateral oophorectomy; or 2. Has not been naturally postmenopausal for at least 24 consecutive months (ie, has had menses at any time in the preceding 24 consecutive months or 730 days.)
    * Conception while on treatment must be avoided.
13. Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy. Prior history of vasectomy does NOT replace requirement for contraceptive use.
14. Subjects must either possess or undergo placement of central venous catheter, including pheresis or trifusion catheter, PICC line, or port.

Exclusion Criteria:

Part One:

1. Prior therapy with anthracycline or checkpoint inhibitors.
2. Hypersensitivity to doxorubicin or any excipients.
3. Patients may not be receiving any other investigational agents (within 4 weeks prior to Cycle 1, Day 1).
4. Prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to Cycle 1, Day 1 or has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
5. Patient has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to Cycle 1, Day 1 or has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier. Subjects with ≤ Grade 2 neuropathy or alopecia are an exception to this criterion and may qualify for the study. Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
6. Additional known malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin, or squamous cell carcinoma of the skin that has undergone potentially curative therapy, or in situ cervical cancer.
7. Patients with underlying immune deficiency, chronic infections including HIV, hepatitis, or tuberculosis (TB) or autoimmune disease.
8. Patients with underlying hematologic issues including bleeding diathesis, such as known previous GI bleeding requiring intervention within the past 6 months. Newly diagnosed pulmonary emboli or deep venous thrombosis must be clinically stable on anticoagulation regimen for ≥ 2 weeks as of Cycle 1 Day 1.
9. Has known history of non-infectious pneumonitis that required oral corticosteroid therapy for resolution within 12 months prior to study entry, or evidence by imaging or symptoms of active non-infectious pneumonitis.
10. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis or leptomeningeal disease. Subjects with previously treated brain metastases may participate provided they are stable based on the following: 1) MRI brain obtained during screening evaluations shows no radiographic evidence of progression or new lesions, 2) any neurologic symptoms have returned to baseline, 3) no requirement for steroids for at least 28 days prior to trial treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability. Patients without a known history of brain metastases do not require screening brain MRI prior to study enrollment.
11. Has received a live vaccine within 30 days of planned start of study therapy. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.
12. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
13. Any uncontrolled, intercurrent illness including but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia
14. Prolonged QTc interval on Screening EKG >475 ms.
15. Ejection Fraction <50% by 2D ECHO at Screening.
16. Any serious medical or psychiatric illness/condition including substance use disorders likely in the judgment of the Investigator(s) to interfere or limit compliance with study requirements/treatment, including NYHA Class II or greater heart disease (see Appendix C for definitions).
17. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
18. Had a previous severe hypersensitivity reaction to another monoclonal antibody.
19. Primary or secondary immunodeficiency (including immunosuppressive disease, autoimmune disease [excluding hypothyroidism, insulin dependent diabetes mellitus, or vitiligo], or usage of immunosuppressive medications).

Part Two: An individual who meets any of the following criteria will be excluded from participation in this study:

1. Prior therapy with anthracycline or checkpoint inhibitors.
2. Hypersensitivity to doxorubicin or any excipients.
3. Patients may not be receiving any other investigational agents (within 4 weeks prior to Cycle 1, Day 1).
4. Prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to Cycle 1, Day 1 or has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
5. Patient has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to Cycle 1, Day 1 or has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier. Subjects with ≤ Grade 2 neuropathy or alopecia are an exception to this criterion and may qualify for the study. Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
6. Additional known malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin, or squamous cell carcinoma of the skin that has undergone potentially curative therapy, or in situ cervical cancer.
7. Patients with underlying immune deficiency, chronic infections including HIV, hepatitis, or tuberculosis (TB) or autoimmune disease.
8. Patients with underlying hematologic issues including bleeding diathesis, such as known previous GI bleeding requiring intervention within the past 6 months. Newly diagnosed pulmonary emboli or deep venous thrombosis must be clinically stable on anticoagulation regimen for ≥ 2 weeks as of Cycle 1 Day 1.
9. Has known history of non-infectious pneumonitis that required oral corticosteroid therapy for resolution within 12 months prior to study entry, or evidence by imaging or symptoms of active non-infectious pneumonitis.
10. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis or leptomeningeal disease. Subjects with previously treated brain metastases may participate provided they are stable based on the following: 1) MRI brain obtained during screening evaluations shows no radiographic evidence of progression or new lesions, 2) any neurologic symptoms have returned to baseline, 3) no requirement for steroids for at least 28 days prior to trial treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability. Patients without a known history of brain metastases do not require screening brain MRI prior to study enrollment.
11. Has received a live vaccine within 30 days of planned start of study therapy. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.
12. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
13. Any uncontrolled, intercurrent illness including but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia
14. Prolonged QTc interval on Screening EKG >475 ms.
15. Ejection Fraction <50% by 2D ECHO at Screening.
16. Any serious medical or psychiatric illness/condition including substance use disorders likely in the judgment of the Investigator(s) to interfere or limit compliance with study requirements/treatment, including NYHA Class II or greater heart disease (see Appendix C for definitions).
17. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
18. Had a previous severe hypersensitivity reaction to another monoclonal antibody.
19. Primary or secondary immunodeficiency (including immunosuppressive disease, autoimmune disease [excluding hypothyroidism, insulin dependent diabetes mellitus, or vitiligo], or usage of immunosuppressive medications).

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2020-01-28 (Actual); Primary Completion 2027-04-07 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Determine the progression-free survival rate | 6 months
  Determine the progression-free survival rate at 6 months of combination therapy with doxorubicin, AGEN1884, and AGEN2034 in anthracycline-naïve patients with advanced or metastatic soft tissue sarcomas.

SECONDARY OUTCOMES:
Determine the overall response rate | 3 years
  Determine the overall response rate of combination therapy with doxorubicin, AGEN1884, and AGEN2034 in anthracycline-naïve patients with advanced or metastatic soft tissue sarcomas.
Determine the clinical benefit rate | 3 years
  Determine the clinical benefit rate of combination therapy with doxorubicin, AGEN1884, and AGEN2034 in anthracycline-naïve patients with advanced or metastatic soft tissue sarcomas.
Determine the duration of response | 3 years
  Determine the duration of response of combination therapy with doxorubicin, AGEN1884, and AGEN2034 in anthracycline-naïve patients with advanced or metastatic soft tissue sarcomas.
Determine the incidence of adverse events | 3 years
  Determine adverse events occurring with combination therapy of doxorubicin, AGEN1884, and AGEN2034 in anthracycline-naïve patients with advanced or metastatic soft tissue sarcomas.

OTHER OUTCOMES:
Measure changes in tumor-infiltrating and circulating immune cells | 3 years
  To measure the change in proportion of various immune cells in tumor biopsies and peripheral blood samples and correlate with response outcomes as a result of combination therapy with doxorubicin, AGEN1884, and AGEN2034 in anthracycline-naïve patients with advanced or metastatic soft tissue sarcomas.

CONTACTS AND LOCATIONS:
Overall Officials: Breelyn Wilky, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Hospital, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No